CLINICAL TRIAL: NCT07211373
Title: Advancing Student Suicide Interventions With Scalable Technologies (ASSIST)
Brief Title: Advancing Student Suicide Interventions With Scalable Technologies
Acronym: ASSIST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of Wisconsin, Madison (Other); University of Massachusetts Chan Medical School, Worcester (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMassIRB6366; P50MH129701 (NIH)
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Suicidal Ideation; Suicide Attempt; Self-Harm
Keywords: suicide; self-harm; attempt; ideation; suicidal thought; suicidal plan; crisis intervention; suicide prevention; emotional support; mental health; behavioral health; technology; mobile application; lethal means; safety plan
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior; Suicide; Suicide Prevention; Psychological Well-Being | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Jaspr (Experimental): Subjects in this arm will complete a guided Safety Planning, and Lethal means counseling on the Jaspr app before open access to the Jaspr resource library.
  Subjects can sign up to receive Jaspr At Home (JAH) mobile app. Subjects will have continue to have access to treatment as usual through their respective university clinics.
  Interventions: Device: Jaspr
- Jaspr+ (Experimental): Subjects in this arm will complete a guided Safety Planning, and Lethal means counseling on the Jaspr app before open access to the Jaspr resource library. This will be guided by motivational interviewing principles.
  Subjects can sign up to receive Jaspr At Home (JAH0 mobile app. Subjects will be prompted with their personalized goals as reminders to use the Jaspr at home app.
  Subjects will have continue to have access to treatment as usual through their respective university clinics.
  Interventions: Device: Jaspr; Behavioral: Behavioral support

INTERVENTIONS:
Device: Jaspr — With assistance from a research staff, the subject will complete self-administered suicide risk assessment on the tablet via Jaspr app, then the subject will engage with suicide-related coping skills and resources that the app provides. Subjects will continue to have access to the coping skills and videos via a mobile app.
Behavioral: Behavioral support — Jaspr conversations will be augmented human-driven behavioral support. Conversations will be guided by motivational interviewing principles. Subjects can sign up to receive JAH mobile app.
  Subjects will be prompted with their personalized goals as reminders to use the Jaspr app.
  Arms: Jaspr+

SUMMARY:
Mobile-based applications, such as JasprHealth, can deliver evidence-based skills intended to reduce imminent suicide risk (e.g., reducing means access), improve emotional states (e.g., via distraction and coaching to act opposite to emotions), and reduce feelings of social isolation (e.g., via shared stories), but user engagement is a barrier. The aim of this study was to examine the effects of a technological application resource (Jaspr) relative to human augmentation (Jaspr+, e.g., motivationally focused orientation plus prompts) on acceptability, preliminary effectiveness, and engagement among college students who screen positive for suicide risk.

DETAILED DESCRIPTION:
Mobile-based applications, such as Jaspr Health, can deliver evidence-based skills intended to reduce imminent suicide risk (e.g., reducing means access), improve emotional states (e.g., via distraction and coaching to act opposite to emotions), and reduce feelings of social isolation (e.g., via shared stories). Although mobile-device-delivered interventions hold the potential to make interventions widely accessible, user engagement presents a substantial barrier to efficacy. This study, ASSIST: Advancing Student Suicide Interventions with Scalable Technologies, aims to improve engagement with mobile-delivered suicide prevention applications, with the ultimate goal of reducing suicidal thoughts and behaviors in college students. Including human elements alongside Jaspr Health has the potential to improve the uptake of this evidence-based, accessible mobile-device-delivered intervention.

The aim of this study was is to examine the effects of the technological application resource Jaspr tablet application with access to Jaspr at Home (JAH) vs. Jaspr+ human augmentation (e.g., motivationally focused orientation plus prompts) on acceptability, preliminary effectiveness, and engagement among 50 college students who screen positive for suicide risk (n=25 per condition) over the course of 2 months. Candidate mechanisms (e.g., coping skills, self-stigma) will also be assessed. Participants were randomized via the Redcap randomization module, stratified by site.

ELIGIBILITY:
Inclusion Criteria:

* Recent suicidal thoughts or behavior (i.e., past 2-week suicidal ideation or past 6-month suicidal behaviors)
* Current UMass Amherst or University of Wisconsin Madison undergraduate student
* 18 years of age or older
* Ability to understand written or spoken English
* Owning a mobile device
* Ability to understand and consent to study procedures

Exclusion Criteria:

* No recent suicidal thoughts or behaviors (i.e., past 2-week suicidal ideation or past 6-month suicidal behaviors)
* Not a current UMass Amherst or University of Wisconsin Madison undergraduate student
* Under 18 years of age
* Inability to understand written or spoken English
* Does not own a mobile device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation | weeks 0, 4, 8
  Assessed with Suicide Ideation Questionnaire [SIQ], with higher scores reflecting greater past month suicidal ideation.
Suicidal behaviors | weeks 0, 1, 2, 3, 4, 8
  Assessed with the Columbia-Suicide Severity Rating Scale [C-SSRS] self-report screen past week (y = presence /n)

SECONDARY OUTCOMES:
Suicide-related coping | weeks 0, 4, 8
  Assessed with the suicide-related coping scale, [SRCS] with higher scores reflecting a better ability to cope with suicidal thoughts
Ways of coping | weeks 0, 4, 8
  Assessed with the DBT-Ways of Coping Checklist (DBT-WCCL), which yields scales of skills use, general dysfunctional coping, and blaming others, with mean scores of 0-3, with higher levels indicating greater use of those strategies.
Suicide stigma | weeks 0, 4, 8
  Assessed with the personal suicide stigma questionnaire [PSSQ], with higher scores reflecting greater stigma.
Self-reported engagement | weeks 0, 1, 2, 3, 4, 8
  Assessed with item developed for this study, with higher scores reflecting greater engagement in the app.
Acceptability | weeks 0, 4, 8
  Assessed with the Acceptability of Implementation Measure [AIM], with higher scores reflecting whether the intervention is liked, welcomed, or approved.
Satisfaction with Intervention | weeks 0, 4, 8
  Assessed with the Client Satisfaction Questionnaire - 8 [CSQ8], with higher scores reflecting greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The analytic plan and de-identifiable/de-identified data will be shared.
Supporting Information: SAP
Time Frame: Data are expected to be cleaned scored and uploaded by Jan 2028 for at least 7 years.
Access Criteria: Data will be available from the researchers upon request

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Posner, K. (2008). Columbia-Suicide Severity Rating Scale. Research Foundation for Mental Hygiene.
- [Background] Neacsiu AD, Rizvi SL, Vitaliano PP, Lynch TR, Linehan MM. The dialectical behavior therapy ways of coping checklist: development and psychometric properties. J Clin Psychol. 2010 Jun;66(6):563-82. doi: 10.1002/jclp.20685. PMID 20455249
- [Background] Maclean BR, Forrester T, Hawgood J, O'Gorman J, Rimkeviciene J. The Personal Suicide Stigma Questionnaire (PSSQ): Relation to Self-Esteem, Well-Being, and Help-Seeking. Int J Environ Res Public Health. 2023 Feb 21;20(5):3816. doi: 10.3390/ijerph20053816. PMID 36900827
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Kelly PJ, Kyngdon F, Ingram I, Deane FP, Baker AL, Osborne BA. The Client Satisfaction Questionnaire-8: Psychometric properties in a cross-sectional survey of people attending residential substance abuse treatment. Drug Alcohol Rev. 2018 Jan;37(1):79-86. doi: 10.1111/dar.12522. Epub 2017 May 7. PMID 28480521
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Gellatly J, Bower P, Hennessy S, Richards D, Gilbody S, Lovell K. What makes self-help interventions effective in the management of depressive symptoms? Meta-analysis and meta-regression. Psychol Med. 2007 Sep;37(9):1217-28. doi: 10.1017/S0033291707000062. Epub 2007 Feb 19. PMID 17306044

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: ASSIST Protocol and SAP (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT07211373/Prot_SAP_000.pdf